CLINICAL TRIAL: NCT03413202
Title: Effectiveness of Butylphthalide on Dynamic Cerebral Autoregulation in Patients With Large-artery Atherosclerosis Acute Ischemic Stroke(EBCAS)
Brief Title: Effectiveness of Butylphthalide on Dynamic Cerebral Autoregulation in Patients With Acute Ischemic Stroke.
Acronym: EBCAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yi Yang (Other)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EBCAS
Record Dates: First submitted 2018-01-18; First posted 2018-01-29 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Acute Ischemic Stroke
Keywords: butylphthalide(NBP); large-artery atherosclerosis acute ischemic stroke; dynamic Cerebral Autoregulation(dCA)
MeSH Terms: conditions — Ischemic Stroke | interventions — 3-n-butylphthalide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- butylphthalide(NBP) (Experimental): Based on the standard medical care, 25mg of NBP injection, and 100ml of 0.9% saline; NBP capsule
  Interventions: Drug: butylphthalide(NBP)
- placebo (Placebo Comparator): Based on the standard medical care, 100ml of 0.9% saline as the placebo; starch capsule as the placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: butylphthalide(NBP) — Standard medical care is in accordance with China Guideline for the diagnosis and treatment of acute ischemic stroke (2014), including medical care for vital signs, control of temperature, blood pressure and glucose, improving cerebral blood circulation, antiplatelet treatment and nutritional supportive care.In addition, 25mg butylphthalide(NBP) injection, and 100ml 0.9% saline by an independent research nurse, sealed with brown bag in order to make the investigators and patients blinded, infusion for 14 days, then, butylphthalide(NBP) capsule for 76 days.
  Arms: butylphthalide(NBP)
Drug: placebo — Standard medical care is in accordance with China Guideline for the diagnosis and treatment of acute ischemic stroke (2014), including medical care for vital signs, control of temperature, blood pressure and glucose, improving cerebral blood circulation, antiplatelet treatment and nutritional supportive care.In addition, 100ml 0.9% saline by an independent research nurse, sealed with brown bag in order to make the investigators and patients blinded, infusion for 14 days, then, starch capsule for 76 days.
  Arms: placebo

SUMMARY:
This is a randomized, triple-blind, placebo-controlled, multicenter clinical trial. Eligible patients will be randomized into either the butylphthalide (NBP) or placebo group in a 2:1 ratio.The main purpose of this study is to determine whether butylphthalide can improve dynamic Cerebral Autoregulation (dCA) in large-artery atherosclerosis acute ischemic stroke.

DETAILED DESCRIPTION:
Cerebral stroke, the first cause of death in China, seriously affects the health and living of people. Its high incidence, disability, mortality and recurrence rate give a heavy burden on the family, society and country. According to TOAST classification, large-artery atherosclerosis ischemic stroke is one of the most common subtypes, and majority experts demonstrate its dynamic Cerebral Autoregulation (dCA) is impaired in affected hemisphere.

Thrombolytic therapy with intravenous tissue plasminogen activator (tPA), which remains the only therapeutic drug for acute ischemic stroke approved by the US Food and Drug Administration, is limited by the narrow time window of thrombolysis, bleeding complications, or high costs. Other treatment strategies mainly utilize therapeutic agents to prevent or reduce cell damage from ischemia. Butylphthalide (NBP) is a multiple target drug for the treatment of acute mild to moderate ischemic cerebral stroke.

Cerebral autoregulation (CA) is the main mechanism that maintains relatively constant cerebral blood flow, which is critical for the normal functioning of physiological functions, as well as the occurrence, development and prognosis of the cerebral stroke.whether NBP can improve the dCA in large-artery atherosclerosis acute ischemic stroke has not been illustrated.

Thus, in this study, investigators plan to enroll 99 eligible patients, which will be randomized into either the NBP or placebo group in a 2:1 ratio within 90 days follow-up to explore whether NBP can improve the dCA in large-artery atherosclerosis acute ischemic stroke. DCA measurement will be performed at 0, 14 and 90 days after entering the trial, nurses will collect intravenous blood 6ml 3 times (each time before dCA measurement, the blood samples will be stored for laboratory test). Clinical information and follow-up information will be collected and recorded in case report form (CRF) once signing of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 18 to 80, both genders;
* Within 48 hours symptoms onset;
* According to TOAST classification, diagnosed to be large-artery atherosclerosis ischemic stroke, without history of stroke in the past three months;
* 5≤National Institutes of Health Stroke Scale (NIHSS) ≤25;
* Unilateral internal carotid artery (ICA) or M1 segment of middle cerebral artery (MCA) stenosis (rate of stenosis ranging from 50-99%);
* Sufficient bilateral temporal bone windows for insonation of the middle cerebral artery;
* Glasgow Coma Scale (GCS) ≥ 8;
* Willing to participate and sign the informed consent.

Exclusion Criteria:

* Patients who have received or plan to undergo intravascular interventional treatment/thrombolytic therapy;
* Coma or agitation, and can't cooperate to complete dCA;
* Has been given butylphthalide injection or capsules;
* Arrhythmia, anemia and hyperthyroidism which may influence the stability of cerebral blood flow diagnosed by two physicians by electrocardiogram and laboratory tests;
* Other intracranial diseases, including cerebral hemorrhage (primary or secondary), intracranial neoplasm, aneurysm, arteriovenous malformation, etc;
* Alanine transaminase (ALT) or glutamic-oxalacetic transaminase (AST) continued to rise more than 3 times the upper limit of normal , creatinine clearance rate<30ml/min;
* Pre-stroke Modified Rankin Scale (mRS) score ≥ 2;
* Malignant neoplasm and expected lifetime < 2 years;
* Pregnant and lactating women;
* Participating in other trials or has been participated in other trials in recent 3 months;
* Dementia and mental illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Phase difference (PD) in degree | within 14 days injection NBP,and 90 days of sequential therapy
  A dCA parameter derived from transfer function analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, MD, PhD, Study Chair — Neuroscience Center, Department of Neurology, The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Derived] Guo ZN, Yue BH, Fan L, Liu J, Zhu Y, Zhao Y, Zhong J, Lou Z, Liu XL, Abuduxukuer R, Zhang P, Qu Y, Shen Z, Shi B, Zhang KJ, Liu J, Chang J, Jin H, Sun X, Yang Y. Effectiveness of butylphthalide on cerebral autoregulation in ischemic stroke patients with large artery atherosclerosis (EBCAS study): A randomized, controlled, multicenter trial. J Cereb Blood Flow Metab. 2023 Oct;43(10):1702-1712. doi: 10.1177/0271678X231168507. Epub 2023 Apr 6. PMID 37021629